CLINICAL TRIAL: NCT07373223
Title: VR-STEM: Virtual Reality Schema Therapy Exercises With Parent and Child Modes
Brief Title: Virtual Reality Schema Therapy Exercises With Parent and Child Modes
Acronym: VR-STEM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22811
Record Dates: First submitted 2025-09-08; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Psychiatric Disorders
Keywords: Virtual Reality Schema Therapy
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: Explorative, non-randomized pilot study with pre-post design (N=30)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VR Schema Therapy Chairwork Exercise (Other): The intervention consists of a schema therapy chairwork exercise in Virtual Reality
  Interventions: Behavioral: VR Schema Therapy Chairwork Exercise

INTERVENTIONS:
Behavioral: VR Schema Therapy Chairwork Exercise — VR Schema Therapy chairwork exercise

SUMMARY:
The goal of this clinical trial is to develop a Virtual Reality version of a Schema Therapy exercise and test its feasibility, acceptability and potential usefulness in people with psychiatric disorders (age 18-65). The main questions the investigators aim to answer are:

1. Are dialogue exercises with virtual reality mode avatars feasible, acceptable and useful?
2. How do patients experience VR schema therapy exercises (in terms of immersion, elicited emotions, therapeutic relationship or subjective efficacy) and are the exercises potentially effective (in terms of schema mode scores, self-criticism, self-compassion and self-esteem)?
3. In case of a potential 'effect', is this moderated by mental imagery ability?

The investigators hypothesize that 1) dialogue exercises with virtual reality mode avatars are feasible, ac-ceptable and useful according the Technology Acceptance Model (TAM; Davis, 1989); 2) patients experience high levels of immersion, elicited emotions and subjective efficacy, a strong therapeutic relationship, and show effects on schema mode scores and self-compassion and self-esteem scores; and 3) these effects are moderated by patients' mental imagery ability in such a way that patients with less mental imagery abilities benefit most.

The development of the VR version of the exercise will be done in collaboration with patients and therapists.

To test its feasibility, acceptability and potential usefulness, participants will be invited to receive one session of the exercise. During this session, they will complete some questionnaires before and after the exercise, and they will be asked about their opinions about and experiences of the exercise.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* In treatment at a tertiary treatment facility (UCP, UMCG)
* Whose current psychological distress is related to early life experiences as indicated by a clinician
* Score of >3 on one of three schema modes on the SMI (Lobbestael et al., 2010)

Exclusion Criteria:

* Insufficient command of the Dutch language
* Primary diagnosis of a substance use disorder, or organic brain disease (such as dementia)
* Unable to provide informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-26 (Estimated); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Screened and enrolled patients per month | From start to end of recruitment (+/- 10 months)
  The amount of screened and enrolled patients per month will be registered to evaluate feasibility and acceptability.
Drop-outs | From start to end of recruitment (+/- 10 months)
  Total number of drop-outs will be registered to evaluate feasibility and acceptability.
Reasons for withdrawal | From start to end of recruitment (+/- 10 months)
  Reasons for withdrawal from the study will be registered to evaluate feasibility and acceptability
Total and types of adverse events | From start to end of recruitment (+/- 10 months)
  The total number and types of adverse events will be registered to evaluate feasibility and acceptability.
Experienced issues during sessions | During the 2-hour sessions (From start to end of recruitment [+/- 10 months])
  Experienced issues during sessions will be registered to evaluate feasibility and acceptability
Evaluative questions | At the end of the 2-hour intervention session (at post-intervention assessment)
  A questionnaire based on the Technology Acceptance Model (TAM) will be completed by patients to evaluate their feedback, perceived usefulness, the added value, and their attitude towards VR schema therapy. This measure is used to evaluate feasibility and acceptability. It consists of 16 questions, divided into two subsections: subjective experience (8 questions) and Technology Acceptance Model (TAM) (8 questions). Questions are scored on a Likert scale ranging from 1 to 7 (total min. 16, max. 112; per subsection min. 8, max. 56). A lower score means a lower evaluation/more negative experience of the intervention, and a higher score means a higher evaluation/more positive experience with the intervention.
Patients qualitative first experiences | At the end of the 2-hour intervention session, after the post-intervention assessment
  Patients qualitative first experiences with the Virtual Reality intervention will be measured using a qualitative, semi-structured interview at the end of each session, to evaluate feasibility and acceptability. Standard questions are:
  1. How did you find the exercise?
  2. What did you find positive about the exercise? (how can we make the positive aspects even more positive?)
  3. What is missing from the exercise? (what can we improve?) The questions are intended as a guiding structure rather than a fixed questionnaire, and allow for additional follow-up questions to explore relevant topics further.

SECONDARY OUTCOMES:
Momentary Schema Modes Questionnaire (MSMQ) | At the start (baseline) and at the end of the single session of 2 hours (pre- and post-intervention)
  The Momentary Schema Modes Questionnaire (MSMQ) will be completed by patients during the session. Difference scores will be used for evaluation of preliminary effects. The MSMQ consists of 35 questions measuring the present-moment level of 11 schema modes. The questions are rated on a Visual Analogue Scale ranging from 0-100 (total min. 0, max. 3500). Lower scores represent a lower presence of a certain schema mode.
Visual Analogue Scales | At the start (baseline) and at the end of the single session of 2 hours (pre- and post-intervention)
  Visual Analogue Scales will be used to measure affect and self-esteem. The questionnaire is derived from previous ESM studies, and consists of 12 questions divided over 3 subscales: positive affect (3 questions), negative affect (3 questions), self-esteem (6 questions). Each question is scored on a scale ranging from 0-100. Difference scores for each subscale are used to evaluate preliminary effects. Higher scores represent higher levels of the measured variable (positive affect [min. 0, max. 300], negative affect [min. 0, max. 300], self-esteem [min. 0, max. 600]).
Self-Compassion and self-Criticism Scales (SCCS) | At the start (baseline) and at the end of the single session of 2 hours (pre- and post-intervention)
  The Self-Compassion and self-Criticism Scales (SCCS) is a questionnaire that measures levels of self-criticism and self-compassion. It consists of 5 situations, for which participants have to score to what extent they would respond to themselves in a reassuring, soothing, contemptuous, compassionate, critical, and harsh way. For the current study, each of the reactions is scored on a Visual Analogue Scale ranging from 0-100 (Self-criticism scale min. 0, max. 1500; self-compassion scale min. 0, max. 1500). Higher scores on the self-criticism scale represent higher levels of self-criticism, whereas higher scores on the self-compassion scale represent higher levels of self-compassion. Difference scores for each scale will be used to evaluate preliminary effects.
Immersion | At the end of the 2-hour intervention session (at post-intervention assessment)
  Two questions from the Igroup Presence Questionnaire (IPQ) will be used to assess immersion into Virtual Reality (VR). Both questions are scored on a Visual Analogue Scale ranging from 0-100 (total min. score 0, max. 200). Lower scores represent lower levels of immersion into the VR environment.
Therapeutic relationship | At the end of the 2-hour intervention session (post-intervention asessment)
  The Session Rating Scale (SRS) will be used to assess working alliance/therapeutic relationship. The SRS consists of 4 questions which are scored on a Visual Analogue Scale ranging from 0-100 (total min. 0, max. 400). Lower scores represent lower levels of experienced therapeutic relationship/working alliance during the intervention session.

OTHER OUTCOMES:
Vividness of Visual Imagery Questionnaire (VVIQ) | At the start of the single intervention session of 2 hours (pre-intervention assessment)
  The Vividness of Visual Imagery Questionnaire (VVIQ) consists of 16 items assessing mental imagery ability. Each question is scored on a Likert scale ranging from 1 to 5, where higher scores represent lower ability of mental imagery. For purposes of interpretation, the scale is recoded in the current study, so that higher scores represent a higher ability of mental imagery.
Visualizer-Verbalizer Questionnaire (VVQ) | At the start of the single intervention session of 2 hours (pre-intervention assessment)
  The Visualizer-Verbalizer Questionnaire (VVQ) consists of 30 items used in this study to assess mental imagery ability. The 30 items are divided over 3 subscales (10 items per subscale), namely visual, verbal, and dream items. These items measure a preference for either a visual or verbal learning style, and vividness of dreams. A more visual learning style and higher vividness of dreams is associated with mental imagery ability. Each question is scored on a binary scale choosing whether a statement is true or false for them. Total scores for each subscale are calculated (min. 0, max. 10), to assess the participants preference for either a visual or verbal learning style, and vividness of dreams. Higher scores represent a higher preference for a learning style or higher vividness of dreams.
Schema Mode Inventory (SMI) | Screening before start of intervention (+/- 1 week before)
  The Schema Mode Inventory (SMI) will be used to screen participants for participation in the study. The SMI consists of 118 items assessing levels of presence of 14 schema modes. Questions are scored on a Likert scale ranging from 1 (never or almost never) to 6 (always). Mean scores are calculated for each schema mode (min. 1, max. 6). A score of >3 on one of three schema modes (demanding parent, punitive parent, and/or vulnerable child) is used as a cut-off for inclusion in the study. Higher levels on the schema modes represent a higher level of presence of the schema mode.
Young Schema Questionnaire - Short Form version 3 (YSQ-SF) | At the start of the single intervention session of 2 hours (at pre-intervention; baseline)
  The Young Schema Questionnaire - Short Form version 3 (YSQ-SF) will be used to assess schemas (core self-beliefs). The YSQ-SF consists of 90 statements (assessing 18 schemas, 5 questions each) which participants rate to what extent the statement is true for them (Likert scale 1 to 6). Mean scores are calculated for each schema (min. 1, max. 6). Higher scores represent a stronger presence of a schema.
Age | At the start of the single intervention session of 2 hours (at pre-intervention; baseline)
  Age in years (min. 18, max. 65)
Biological sex | At the start of the single intervention session of 2 hours (at pre-intervention; baseline)
  Biological sex
Education | At the start of the single intervention session of 2 hours (at pre-intervention; baseline)
  Educational level of the participant (highest completed)
Working status | At the start of the single intervention session of 2 hours (at pre-intervention; baseline)
  Working status; (employed, looking for a job [unemployed], student, receiving benefits, other)
Living situation | At the start of the single intervention session of 2 hours (at pre-intervention; baseline)
  Living situation, possible options: alone, with partner, with family/parents, supported/assisted living, other
Diagnosis | At the start of the single intervention session of 2 hours (at pre-intervention; baseline)
  Primary diagnosis (according to the Diagnostic and Statistical Manual of mental disorders, 5th edition [DSM-5]). Open-ended question.
Illness duration | At the start of the single intervention session of 2 hours (at pre-intervention; baseline)
  Illness duration (in years and months)
Previous psychological treatment | At the start of the single intervention session of 2 hours (at pre-intervention; baseline)
  Previous received psychological treatment (Psychological treatment, inpatient psychiatric hospitalization, and/or day treatment)
Current psychological treatment | At the start of the single intervention session of 2 hours (at pre-intervention; baseline)
  Currently receiving psychological treatment (Yes/no, if yes: type, duration and frequency)
Current medication | At the start of the single intervention session of 2 hours (at pre-intervention; baseline)
  Currently taking any medication (yes/no, if yes: type and dosage)

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Centre Groningen, Groningen, Provincie Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon reasonable request after publication of the manuscript
Time Frame: Upon publication of the manuscript
Access Criteria: Data will be shared upon reasonable request after publication of the manuscript